CLINICAL TRIAL: NCT03839836
Title: Variation of Spatiotemporal Parameters in School Children Carrying Different Backpack Loads: Clinical Trial
Brief Title: Variation of Spatiotemporal Parameters in School Children Carrying Different Backpack Loads
Acronym: SCBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Gabriel Gijon-Nogueron, Assistant Professor, University of Malaga
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: UMalagaHS
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Child, Only; Gait, Unsteady
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Clinical trial experimental
Who Masked: Participant, Investigator
Masking Description: The study was a double-blind, five-arm experimental study. This biomechanical study was designed to examine the effect of weight in the gait of the children with the backpack, no follow-up was undertaken.
  A convenience sample of children was approached The potential recruits are asked to attend a screening appointment Children were asked to walk naturally, facing forward, with their hands out of pockets; wearing light, comfortable clothes, with the BP placed correctly with 5 different weights inside the backpack.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Baseline (No Intervention): Children between six and 12 years, no pain in the lower limb and back at the time of examination using a backpack without the child's body weight, the spatio-temporal parameters are measured with the OptoGait® system
- 5% child's body weight (Experimental): Children between six and 12 years, no pain in the lower limb and back at the time of examination using a backpack load was added to the BPs 5%, of the child's body weight, the spatio-temporal parameters are measured with the OptoGait® system
  Interventions: Other: Backpack child's body weight
- 10% child's body weight (Experimental): Children between six and 12 years, no pain in the lower limb and back at the time of examination using a backpack load was added to the BPs 10%, of the child's body weight, the spatio-temporal parameters are measured with the OptoGait® system
  Interventions: Other: Backpack child's body weight
- 15% child's body weight (Experimental): Children between six and 12 years, no pain in the lower limb and back at the time of examination using a backpack load was added to the BPs 15%, of the child's body weight, the spatio-temporal parameters are measured with the OptoGait® system
  Interventions: Other: Backpack child's body weight
- 20% child's body weight (Experimental): Children between six and 12 years, no pain in the lower limb and back at the time of examination using a backpack load was added to the BPs 20%, of the child's body weight, the spatio-temporal parameters are measured with the OptoGait® system
  Interventions: Other: Backpack child's body weight

INTERVENTIONS:
Other: Backpack child's body weight — Children are asked to walk naturally, facing forward, with their hands out of pockets; wearing light, comfortable clothes, with the BP placed correctly. As the children start walking, the researchers select the foot of the first step inside the bars, in the Optogait software. After being instructed to 'walk slowly at a comfortable speed', the children walk from a point two metres in front of the bar and stop at a point two metres behind the last bar, to minimize effects of acceleration and deceleration . A three-minute interval occurs between individual assessments to transmit the data, as well as to prepare for the next assessment. Only steps in the sensor areas are included in the analysis. Recording six to eight strides is reported as sufficient to obtain representative data for unimpaired adults. Subsequently, five experimental conditions are measured: without BP, BP loads of 5%, 10%, 15%, and 20% of body weight. The order of these loaded conditions are random.
  Arms: 10% child's body weight; 15% child's body weight; 20% child's body weight; 5% child's body weight

SUMMARY:
Backpacks (BP) represent the method most used by students to transport external cargo. Previous studies cite that between 4.7% and 38% of children carry daily BP loads greater than 20% of their body mass. The purpose of this study was to analyze spatiotemporal parameters of gait in children using varyingly loaded BPs.

DETAILED DESCRIPTION:
This study examined 231 schoolchildren (118 boys, 113 girls) aged six to 12 years, carrying a traditional BP to manipulate loading (Crossing Backpack Children Arpenaz 7 Litres, Junior Red Quechua). The inclusion criteria were: age between six and 12 years, no pain in the lower limb and back at the time of examination. The exclusion criteria were: recent injury to the lower limb and back, alterations in the foot bones, congenital structural changes to the ankle, flatfoot associated with cerebral palsy, surgical treatment of foot or lower leg, or any genetic, neurologic or muscular conditions.

The parents were provided with information about the study, and those consenting for their children to participate, also completed a questionnaire. The children were fully informed of the procedures involved and gave assent. All procedures were in accordance with the ethical standards of the institution of University of Malaga (CEUMA 91/2016H) and with the 1964 Helsinki declaration.

Load was added to the BPs in increments of 5%, 10%, 15% and 20% of the child's body weight. Spatio-temporal parameters were measured with the OptoGait® system.

Two examiners were responsible for the system software and collecting data. General information, including height and weight, were recorded. To measure gait parameters, the protocol used for the Optogait reliability testing was used. This involved the children walking on a walkway at a comfortable speed, repeating this walk three times and calculating the mean speed. Prior to data collection, the children performed one familiarization trial for five minutes. Children were asked to walk naturally, facing forward, with their hands out of pockets; wearing light, comfortable clothes, with the BP placed correctly. As the children started walking, the researchers selected the foot of the first step inside the bars, in the Optogait software. After being instructed to 'walk slowly at a comfortable speed', the children walked from a point two metres in front of the bar and stopped at a point two metres behind the last bar, to minimize effects of acceleration and deceleration

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were: age between six and 12 years, no pain in the lower limb and back at the time of examination.

Exclusion Criteria:

* The exclusion criteria were: recent injury to the lower limb and back, alterations in the foot bones, congenital structural changes to the ankle, flatfoot associated with cerebral palsy, surgical treatment of foot or lower leg, or any genetic, neurologic or muscular conditions.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — 6 to 12 years
Enrollment: 231 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
OptoGait® system is a system for movement analysis and functional assessment of patients with five-meter instrument walkway test | 1 hour
  The Optogait is a reliable and validated system, which records 19 spatio-temporal parameters. For this study, a five-metre instrument walkway is used, consisting of five transmission bars and five reception bars, with a separation of 120cm. Each bar (100cm x 8cm) contains 96 light emitters 3mm from the ground. Optical sensors operate at a frequency of 1000 Hz, with accuracy of 1cm, to detect the spatio-temporal parameters related to walking, running and other movements. The software use is OptoGait® v.1.11.1.0. The Optogait system is calibrated and checked for accuracy at all times, and provided an exhaustive, reliable measurement of the spatiotemporal phases of the gait cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriel Gijon Nogueron, Armilla, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paez-Moguer J, Montes-Alguacil J, Garcia-Paya I, Medina-Alcantara M, Evans AM, Gijon-Nogueron G. Variation of spatiotemporal parameters in school children carrying different backpack loads: a cross sectional study. Sci Rep. 2019 Aug 21;9(1):12192. doi: 10.1038/s41598-019-48675-3. PMID 31434980